CLINICAL TRIAL: NCT06095037
Title: Examining the Effectiveness of Mindful Yoga in Enhancing Psychological Well-being Among Older Adults Discharged From Hospital and Their Caregivers: A Cluster Randomized Controlled Trial
Brief Title: Mindful Yoga for Older Adults and Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Xiaochen Zhou, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Mindfulyoga
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mindful yoga
  Interventions: Behavioral: Mindful yoga
- Control (Active Comparator): Psychoeducation
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindful yoga — 12 week mindful yoga intervention
  Arms: Intervention
Behavioral: Psychoeducation — 12 week psychoeducation sessions
  Arms: Control

SUMMARY:
This study will adopt the intervention of mindful yoga to improve the psychological well-being of older adults who discharged from hospital and their caregivers in Hong Kong.

DETAILED DESCRIPTION:
In the proposed study, the investigators will conduct a fully powered, double-blind, and multicentered randomized controlled trial (RCT) of the efficacy of mindful yoga versus a psychoeducation control. The study sample will consist of older adults discharged from hospitals within the previous 3 months and their informal caregivers. The investigators will aim to determine: (1) the efficacy of mindful yoga in the study group versus the control group in improving the dyadic psychological well-being (as measured by depression, anxiety, stress, and meaning of life) of older adult-caregiver dyads (e.g., both actor and partner effects); (2) whether these improvements were maintained after 3 and 6 months; and (3) the lived experiences of older adults and their caregivers. The investigators hypothesize that: (1) mindful yoga will be more efficacious in improving outcomes compared with the control condition; (2) there will be both actor and partner effects of the intervention on the primary and secondary outcomes; and (3) these outcome improvements will be maintained at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Older adults discharged from hospital

* older adults aged 65 years or above;
* individuals who have been discharged from a local hospital within the previous 3 months who qualify for the Pilot Scheme on Support for Elderly Persons Discharged from Public Hospitals after Treatment and are receiving services from community support services;
* individuals with no mobility issues or who have limited mobility but can access the intervention sites using a wheelchair and are capable of practicing mindful yoga, even if in a wheelchair; and
* individuals who can understand Cantonese.

Caregivers:

• living with older adults during the transition period from hospital to home.

Exclusion Criteria:

Older adults discharged from hospital

* older adults diagnosed with depression, anxiety, or stress disorders by certified doctors;
* older adults diagnosed with severe dementia;
* homebound older adults who face difficulty attending the intervention sites; and
* older adults having a tech-enabled Hospital Admission Risk Reduction Program for the Elderly (HARRPE) score <0.17 or >0.29.

Caregivers:

• Family caregivers who have been diagnosed with severe mental health issues will be excluded from the proposed study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
The Depression, Anxiety, and Stress Scale | Through study completion, an average of 12 weeks
  The total score ranges from 0 to 63. Higher score indicates higher level of depression, anxiety and stress

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire | Through study completion, an average of 12 weeks
  The total score ranges from 39 to 195. Highers score indicates higehr level of mindfulness
Five Facet Mindfulness Questionnaire | 3 months follow-up
  The total score ranges from 39 to 195. Highers score indicates higehr level of mindfulness
Five Facet Mindfulness Questionnaire | 6 months follow-up
  The total score ranges from 39 to 195. Highers score indicates higehr level of mindfulness
The meaning in life scale | Through study completion, an average of 12 weeks
  The total score ranges from 10 to 70. Higher scores indicates higher level of meaning in life
The meaning in life scale | 3 months follow-up
  The total score ranges from 10 to 70. Higher scores indicates higher level of meaning in life
The meaning in life scale | 6 months follow-up
  The total score ranges from 10 to 70. Higher scores indicates higher level of meaning in life
The Depression, Anxiety, and Stress Scale | 3 months follow-up
  The total score ranges from 0 to 63. Higher score indicates higher level of depression, anxiety and stress
The Depression, Anxiety, and Stress Scale | 6 months follow-up
  The total score ranges from 0 to 63. Higher score indicates higher level of depression, anxiety and stress

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wang, Principal Investigator — Lingnan University
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data without participants' privacy information will be shared
Supporting Information: Study Protocol, SAP
Time Frame: The supporting documents will be shared June 30, 2024
Access Criteria: Anyone can access to the supporting documents